CLINICAL TRIAL: NCT05966493
Title: A Randomized, Multicenter, Double-Masked, Vehicle-Controlled Phase 2 Study to Evaluate the Safety and Efficacy of NEXAGON® (Lufepirsen Ophthalmic Gel) in Subjects With Persistent Corneal Epithelial Defects (NEXPEDE-1)
Brief Title: A Study to Evaluate the Safety and Efficacy of NEXAGON® (Lufepirsen Ophthalmic Gel) in Subjects With PCED
Acronym: NEXPEDE-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLK-601-01 (AMB-01-006)
Record Dates: First submitted 2023-06-20; First posted 2023-07-28 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Persistent Corneal Epithelial Defect
Keywords: PCED; Corneal Defect; PED

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NEXAGON® (lufepirsen ophthalmic gel) High Dose Concentration (Experimental): Lufepirsen (High dose concentration) applied topically to the eye once a week for a minimum of 4 weeks to a maximum of 8 weeks.
  Interventions: Drug: lufepirsen high dose
- NEXAGON Vehicle (ophthalmic gel) (Placebo Comparator): Vehicle applied topically to the eye once a week for a minimum of 4 weeks to a maximum of 8 weeks.
  Interventions: Drug: Vehicle
- NEXAGON® (lufepirsen ophthalmic gel) Low Dose Concentration (EU sites only) (Experimental): Lufepirsen (Low dose concentration) applied topically to the eye once a week for a minimum of 4 weeks to a maximum of 8 weeks. (EU sites only).
  Interventions: Drug: lufepirsen low dose

INTERVENTIONS:
Drug: lufepirsen high dose — Lufepirsen is an unmodified connexin43 antisense oligonucleotide.
  Other Names: NEXAGON®
  Arms: NEXAGON® (lufepirsen ophthalmic gel) High Dose Concentration
Drug: Vehicle — Matching vehicle without lufepirsen.
  Other Names: Placebo
  Arms: NEXAGON Vehicle (ophthalmic gel)
Drug: lufepirsen low dose — Lufepirsen is an unmodified connexin43 antisense oligonucleotide.
  Other Names: NEXAGON®
  Arms: NEXAGON® (lufepirsen ophthalmic gel) Low Dose Concentration (EU sites only)

SUMMARY:
This study is to evaluate the safety and efficacy of NEXAGON® (lufepirsen ophthalmic gel) (NEXAGON) in subjects with persistent corneal epithelial defects (PCED). The objectives of the study are to evaluate the safety and efficacy of NEXAGON in this population.

DETAILED DESCRIPTION:
This study is a randomized, multicenter, double-masked, vehicle-controlled study to evaluate the safety and efficacy of NEXAGON (lufepirsen ophthalmic gel) in subjects with persistent corneal epithelial defects (PCED). The study will enroll subjects who will complete a Screening Period, Treatment Period (up to 8 weeks) and Follow-up Period (4 weeks). Those subjects whose defect has not re-epithelialized by the completion of the Treatment Period or who achieved re-epithelialization but failed to maintain re-epithelialization for 28 days after treatment completion (durability) are eligible to enter the NEXAGON Open-label Treatment Period for an additional 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Have a PCED that is at least 2 weeks in duration and refractory to one or more conventional non-surgical standard of care (SOC) treatments
2. Have no clinical evidence of improvement in the PCED within 2 weeks prior to randomization despite the use of non-surgical SOC treatment
3. Subject must provide written informed consent (or assent)
4. Subjects with childbearing potential must be 1-year postmenopausal, surgically sterilized, or have a negative urine pregnancy test

Exclusion Criteria:

1. Have a known ocular infection that is deemed to be active requiring therapeutic intervention
2. Present with a corneal surface defect in either eye that is directly attributed to an infectious etiology (bacterial, viral, fungal and/or protozoal) that has not fully resolved and/or treatment has not been completed
3. Present with evidence of corneal ulceration/melting involving the posterior third of the stroma and/or perforation in either eye
4. Have a blepharitis or meibomian gland disease in the study eye that is deemed to be clinically relevant and/or active
5. Have a history of ocular surgery or any ocular procedure(s) not meeting the designated washout time
6. Have any other ocular disease requiring topical ocular medication in the affected eye
7. Have a presence or history of any ocular or systemic disorder or condition that could interfere the safety or efficacy of the study treatment, or the interpretation of the study results
8. Have a known hypersensitivity to one of the components of the study or procedural medications (e.g., NEXAGON, fluorescein)
9. Participated in an interventional clinical drug or device trial within 28 days prior to Day 1
10. Use of the medications presented in the protocol that are prohibited in the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Achieve Corneal Re-epithelialization Including Durability (CRC) | End of Study: 28 Days after achieving re-epithelialization
  The proportion of subjects achieving corneal re-epithelialization that is maintained for a minimum of 28 days, based on assessment of corneal fluorescein staining images of the PCED by a Central Reading Center (CRC).

CONTACTS AND LOCATIONS:
Overall Officials: Luis G. Vargas, MD, Study Director — Glaukos Corporation
Locations (27):
- United States (20):
  - Glaukos Investigative Site, Dothan, Alabama
  - Glaukos Investigative Site, Petaluma, California
  - Glaukos Investigative Site, Torrance, California
  - Glaukos Investigative Site, Colorado Springs, Colorado
  - Glaukos Investigative Site, Grand Junction, Colorado
  - Glaukos Investigative Site, Bradenton, Florida
  - Glaukos Investigative Site, Fort Myers, Florida
  - Glaukos Investigative Site, South Miami, Florida
  - Glaukos Investigative Site, Atlanta, Georgia
  - Glaukos Investigative Site, Carmel, Indiana
  - Glaukos Investigative Site, Fraser, Michigan
  - Glaukos Investigative Site, Kansas City, Missouri
  - Glaukos Investigative Site, Palisades Park, New Jersey
  - Glaukos Investigative Site, Shelby, North Carolina
  - Glaukos Investigative Site, Bala-Cynwyd, Pennsylvania
  - Glaukos Investigative Site, Nashville, Tennessee
  - Glaukos Investigative Site, Houston, Texas
  - Glaukos Investigative Site, San Antonio, Texas
  - Glaukos Investigative Site, Madison, Wisconsin
  - Glaukos Investigative Site, Milwaukee, Wisconsin
- Germany (2):
  - Glaukos Investigative Site, Mainz
  - Glaukos Investigative Site, München
- Glaukos investigative Site, Messina, Italy
- Spain (4):
  - Glaukos Investigative Site, Barcelona
  - Glaukos Investigative Site, Madrid
  - Glaukos Investigative Site, Seville
  - Glaukos Investigative Site, Zaragoza

IPD SHARING:
Plan to Share IPD: No